CLINICAL TRIAL: NCT04820933
Title: A Switch Clinical Trial of Antiretrovirals to Compare the Impact of Doravirine Versus Integrase Inhibitors With Backbone of Emtricitabine and Tenofovir Alafenamide on Instigators of Atherosclerosis in Persons With Chronic Treated HIV.
Brief Title: Doravirine Versus Integrase Inhibitors on Backbone of Emtricitabine and Tenofovir Alafenamide in HIV
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Theodoros Kelesidis, Principal Investigator, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MISP# 60720 ; STU-2023-0724
Record Dates: First submitted 2021-03-22; First posted 2021-03-29 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: HIV I Infection; Cardiovascular Risk Factor; Lipid Metabolism Disorders
Keywords: HIV; Antiretroviral therapy; Cardiovascular disease
MeSH Terms: conditions — Lipid Metabolism Disorders; Cardiovascular Diseases | interventions — doravirine; emtricitabine tenofovir alafenamide; Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Doravirine plus emtricitabine and tenofovir alafenamide fumarate (Experimental): PIFELTRO (doravirine) 100 mg tablet one daily for 3 months Descovy (200 mg emtricitabine + 10 mg tenofovir alafenamide fumarate) tablet one daily for 3 months
  Interventions: Drug: Doravirine 100 Mg

INTERVENTIONS:
Drug: Doravirine 100 Mg — Doravirine 100 Mg orally dail
  Other Names: Descovy (200 mg emtricitabine + 10 mg tenofovir alafenamide fumarate)

SUMMARY:
This research application will explore the impact of the Non-nucleoside reverse transcriptase inhibitor (NNRTI) doravirine in the setting of established Nucleoside reverse transcriptase inhibitors (NRTIs) backbone [Tenofovir alafenamide (TAF) / Emtricitabine (FTC) as a possible therapeutic strategy to minimize the detrimental impact of ART-related toxicities on metabolism and instigators of atherosclerosis. Given the possible favorable role of NNRTI in pathogenesis of HIV-related dyslipidemia and cardiovascular disease (CVD), this research will provide mechanistic insights into HIV pathogenesis and safety data regarding doravirine (DOR). These data may promote DOR as a robust "HDL friendly" and "metabolism friendly", therapeutic agent that may attenuate morbidity in chronic treated HIV infection. Towards this aim, the investigators will study DOR-related effects on HDL (HDL-C levels and function) and ex vivo assays that determine key molecular determinants of atherogenesis.

DETAILED DESCRIPTION:
Aim 1: To evaluate the relative in vivo impact of DOR on independent measures of HDL function (antioxidant function, cholesterol efflux) compared to integrase inhibitors (raltegravir, dolutegravir, elvitegravir, bictegravir) in the setting of TAF backbone in HIV infected persons with dyslipidemia.

Aim 2: To evaluate the relative in vivo impact of DOR on ex vivo atherogenesis (monocyte-derived foam cell efflux and chemotaxis) compared to integrase inhibitors (raltegravir, dolutegravir, elvitegravir, bictegravir) in the setting of TAF backbone.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Cases: Chronically infected and on anti-retroviral therapy with suppressed viremia for at least 3 months (viral RNA <50 copies per ml)
* On stable antiretroviral therapy for >6 months with Genvoya (elvitegravir 150 mg/cobicistat 150 mg/emtricitabine 200 mg/tenofovir alafenamide 10 mg; E/C/F/TAF) 2) Biktarvy (bictegravir 50 mg/ emtricitabine 200 mg/tenofovir alafenamide 25 mg; B/F/TAF).
* Dyslipidemia (Defined based on use of lipid lowering medications or abnormal baseline lipids (total cholesterol, triglycerides, high density lipoprotein): Rationale: Enrolling participants with dyslipidemia will determine whether switching from TAF/FTC/integrase inhibitor regimen to TAF/FTC/doravirine regimen will directly improve the lipids over 3 months within the same participant.
* Adequate renal function determined by the Cockcroft-Gault formula for creatinine clearance (>60 mL/min/1.73 m2
* Able and willing to provide written consent

Exclusion Criteria:

* • Pregnancy

  * Hepatitis; no evidence of acute hepatitis in the prior 30 days
  * History of severe renal impairment (eGFR < 30 ml/min/1.73 m2)
  * History of severe or recent cardiac event
  * Current alcoholism or IV drug abuse
  * Use of systemic immunomodulatory medications (e.g. steroids) within 4 weeks of enrollment
  * Anemia precluding safe donation of blood (For men, anemia is typically defined as hemoglobin level of less than 13.5 gram/100 ml and in women as hemoglobin of less than 12.0 gram/100 ml).
  * Use of any investigational products within 4 weeks of enrollment
  * Any other clinical condition or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for the study or unable to comply with the study requirements. Such conditions may include, but are not limited to, current or recent history of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurological, or cerebral disease.
  * Subjects who are on medications that are strong inducers of CYP3A (as these may decrease the efficacy of Stribild or Genvoya). Examples include phenobarbital, phenytoin, carbamazepine, and rifampin.
  * Subjects who are on medications that are cleared by CYP3A and that may be toxic with elevated drug levels (examples include Cisapride, ergotamine, Pimozide, Lurasidone, Lovastatin, and Simvastatin).

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
HDL function | 12 weeks post switch of antivirals
  Primary outcome (instigator of atherosclerosis). This is a measure of the lipid peroxide content of HDL per specific amount of HDL relative to the measure of this value in a pooled healthy control (normalized ratio; no units).
Monocyte chemotaxis | 12 weeks post switch of antivirals
  Primary outcome (instigator of atherosclerosis). This is a measure of the ability of isolated blood monocytes to migrate through a trans endothelial layer in an ex vivo model of atherogenesis. Units are % of monocytes that migrated (% chemotaxis).
Monocyte derived foam cell formation of monocytes | 12 weeks post switch of antivirals
  Primary outcome (instigator of atherosclerosis). This is a measure of the ability of isolated blood monocytes to take up lipids and form foam cells in an ex vivo model of atherogenesis. Units are % of monocytes that became foam cells (% Monocyte derived foam cell formation).

SECONDARY OUTCOMES:
Total cholesterol | 12 weeks post switch of antivirals
  Secondary outcome (instigator of atherosclerosis). Units are mg/dl.

CONTACTS AND LOCATIONS:
Overall Officials: Theodoros Kelesidis, MD PHD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No